CLINICAL TRIAL: NCT04832126
Title: Genetic Analysis of Heart Channelopathies in Brazilian Patients and Their Relatives
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Nilson Araújo de Oliveira Junior, Dr., D'Or Institute for Research and Education
Other Study IDs: PRJ1801
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Channelopathies
Keywords: channelopathies; arrhythmia; genetic analysis; Sudden cardiac death
MeSH Terms: conditions — Channelopathies; Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA is purified from peripheral blood or mouth swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: patients with channelopathies
  Interventions: Genetic: Genetic analysis
- Family: relatives of patients with channelopathies
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — Genomic DNA will be purified from peripheral blood or mouth swabs. Whole blood will be collected by peripheral phlebotomy in tubes containing K2EDTA as an anticoagulant. Blood samples will be stored at 4-8 oC for up to a week before DNA purification. Mouth swabs will be collected using the ORAcollect • DNA kit (OCR-100) (DNA Genotek Inc., Canada). Genomic DNA from whole blood or mouth swab samples will be purified using DNeasy Blood & Tissue Kit (QIAGEN).

SUMMARY:
several genes have been associated with ion channel diseases, but a large number of families do not yet have an identified genetic cause. There is a lack of information on the genetic characteristics of channelopathies in Brazilians affected by these diseases. This study aims to carry out a comprehensive genetic analysis of cardiac channelopathies in Brazilian patients and their families. The study will involve 20 patients and 80 family members (a total of 100 individuals) accompanied by the Rede D'Or arrhythmia group in Rio de Janeiro. Individuals will be recruited and subjected to DNA sequencing and phenotypic evaluation, including clinical evaluation, echocardiography, 24-hour Holter or longer electrocardiographic monitoring. An integrated analysis of phenotype-genotype will be made in all individuals included in the study. Patients and their families will be followed up annually for 2 to 5 years through clinical evaluations and the same complementary methods described. The DNA sequencing of patients and their families may contribute to improve the diagnosis of channelopathies and allow the determination of the pattern of occurrence of the disease in the cases involved. Besides, this study may lead to the discovery of new genetic variants associated with channelopathies that will serve as a basis for designing and carrying out broader molecular epidemiological studies. The study of the molecular genetics of channelopathies is important mainly so that patients can avoid sudden death, but also for the medical community, researchers, laboratories, companies involved in the production of medical devices, and public health authorities

DETAILED DESCRIPTION:
Inherited arrhythmias are characterized by variable expressiveness and incomplete penetrance. Extensive genotype-phenotype studies are needed to elucidate the genetic basis of these diseases. There are several reasons for studying the molecular genetics of channelopathies, such as determining the molecular epidemiology of these diseases, offering evidence for a better understanding of the molecular basis of diseases, determining the genetic patterns of occurrence (inherited or again), and improving the diagnosis and genetic counseling. Besides, the genetic study of these diseases can lead to the discovery of new genetic variants associated with these diseases and to the creation of experimental models.

Genetic testing is recommended (Class I) for any patient with a strong clinical suspicion of genetically inherited channelopathies including long QT syndrome, catecholaminergic polymorphic ventricular tachycardia, Brugada syndrome, and short QT syndrome. Specific genetic testing for the mutation identified in the index case is also recommended (Class I) for family members.

The molecular genetics of cardiac channelopathies has been extensively studied in populations in developed countries. In the past, the most frequently used methods were the sequencing of a single or a few suspect genes. More recently, wider panels or even the sequencing of the complete exome have been increasingly used. This procedure has allowed the discovery of an increasing number of genetic variants.

Although the genetic basis for many cases of these diseases is known, many families do not yet have a definite genetic cause. Besides, it is difficult to predict the pathogenicity and clinical evolution of individual mutations. Recent advances in the generation of induced pluripotent stem cells (iPS) may allow considerable progress in the translational research of arrhythmias.

Since the discovery of the first channelopathy in 1995 , the use of genetic tests for diagnostic and prognostic purposes has evolved considerably and is now being used in clinical practice and not just for research purposes. Despite all these advances, the use of DNA sequencing to determine the presence or absence of some diseases is a challenge, since all these clinical syndromes can be associated with different mutations, many of which have not yet been described. The genetic sequencing of patients with genetically inherited arrhythmias is essential not only to provide clinical information related to well-characterized mutations but also to contribute to the discovery of new genetic alterations. In Brugada syndrome, for example, although 12 genotypes have been described so far, genetic changes have been identified in only 30% of cases. The reason for these discrepancies is related to still incomplete knowledge of all the pathways involved in the function and regulation of cardiac ion channels.

Brief descriptions of the most studied channelopathies are presented below. Long QT syndrome (LQTS) This disease has been identified in different areas of the world, in different ethnic groups. Although at least 13 forms of the disease have been described so far, the cause in approximately 20% of cases is not yet defined.

The disease is characterized by a prolongation of the QT interval and arrhythmic events. The arrhythmias usually found in these patients are episodes of polymorphic ventricular tachycardia (torsades de pointes) that causes dizziness and syncope and may progress to ventricular fibrillation and sudden death. Individuals affected by LQTS are more susceptible to atrial fibrillation than the general population This being the most studied channelopathy, the correlation between genetic variants and clinical evolution is very high. Currently, it is known that exercise and emotional stress trigger arrhythmias in patients with LQT1 and that patients with LQT3 usually have episodes of arrhythmia during sleep. It is also known that LQT8 is extremely aggressive with symptoms appearing early and a poor response to treatment. At least 20% of genetically proven LQTS cases have normal ECG. For all these reasons, LQTS is an example of how genetic characterization can help in understanding the pathophysiology of a clinical condition and improve treatment.

Brugada Syndrome (BRS) This clinical syndrome is characterized by spontaneous episodes of polymorphic ventricular tachycardia that can degenerate into ventricular fibrillation and a typical electrocardiographic pattern of elevation of the ST segment from V1 to V3.

The prevalence of this disease is higher in Asia where, in some locations, it is considered the most common cause of natural death among men under 50 years old.

The syndrome usually begins in adulthood, being rare in children. Several genotypes have already been described, typically involving a decrease in the currents of sodium (Na) or an increase in the currents of potassium (K). The pattern of inheritance is autosomal dominant, so half of the family members are expected to be affected. As mentioned earlier for LQTS, the molecular genetics of several cases with clinical criteria for Brugada syndrome has not yet been elucidated.

The treatment of choice is the implantation of a defibrillator. No pharmacological treatment is safe, although isoproterenol or quinidine can be used in cases of electrical storms. Ablation is being investigated to control some of these patients.

The diagnosis is made from the electrocardiogram (ECG) with a typical pattern associated with the clinical evidence of the disease. Occasionally a provocative drug test may be necessary, as the typical pattern may be transient. Blockers of Na channels such as ajmaline can help to identify these patients.

Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT) This disease is characterized by arrhythmic events of bidirectional or polymorphic ventricular tachycardia triggered by an adrenergic stimulus. Baseline ECG and imaging tests are nonspecific. Ventricular arrhythmias are observed exclusively during efforts so that the stress test and the Holter are important diagnostic methods. Two types of mutations have been described so far. One at the ryanodine receptor and the other at the gene encoding calsequestrin. Only 60% of diagnosed individuals carry one of these mutations and, therefore, other genes must be involved. Other conditions Several other arrhythmic genetic syndromes have been described, such as short QT syndrome, sudden unexplained death syndrome, idiopathic ventricular fibrillation, early repolarization, and some genetic forms of atrial fibrillation. Many patients are diagnosed after an episode of sudden aborted death. Better genetic categorization of these cases could help to better understand the mechanisms involved in these diseases and improve treatment. Family screening and adequate genetic counseling are essential.

OBJECTIVES PRIMARY OBJECTIVE This study aims to carry out a comprehensive genetic analysis of cardiac channelopathies in Brazilian patients and their families.

SECONDARY OBJECTIVES Discover new genetic variants that are causal or associated with arrhythmias. Determine the molecular epidemiology of these diseases. Find evidence for a better understanding of the molecular basis of these diseases.

Allow the creation of experimental models. Determine the genetic patterns of occurrence (inherited or new, among others). Allow an improvement in the diagnosis. Enable an improvement in genetic counseling.

HYPOTHESES Genetic analysis will improve the diagnosis and genetic counseling of patients and their families. Early diagnosis can prevent sudden death in some cases. There is a possibility to detect new genetic variants associated with channelopathies.

METHODS STUDY DESIGN AND POPULATION 20 patients and 80 family members (a total of 100 individuals) accompanied by the arrhythmia group of Rede D'Or will be recruited. The total number of individuals to include in the study refers to a convenience sample based on patients currently followed by the group of specialists from Rede D'Or who are part of the study and their families. The choice of up to 4 family members per proband is justified by the fact that this number of related individuals is, in most cases, sufficient to determine the pattern of occurrence and segregation of phenotypes.

The specification of the family members of each proband that will be included will be made on a case-by-case basis depending on the pattern of genetic inheritance, the family composition, and the availability of samples from other family members. The inheritance pattern of causal genetic variants or those associated with phenotypes jointly defined as cardiac channelopathies is, more commonly, autosomal dominant. In this context, the genetic testing of both parents and, whenever possible, of first-degree relatives affected or not by the phenotype is sufficient for the establishment or exclusion of causality. Although less common, sporadic cases can also be seen. In such cases, the pathogenic genetic variant should not be detected in the parents but testing them is necessary to confirm the sporadic pattern. In these cases, siblings and/or first-degree relatives should only be tested in the absence of the parents.

This is a pilot study that will provide information on the population affected by these diseases in our country. All eligible patients, affected by channelopathies and followed up in hospitals and clinics belonging to Rede D'Or São Luiz in Rio de Janeiro and selected family members, will be invited to participate in the study. DNA sequencing will be performed 3 ± 2 months after inclusion. The phenotypic analysis will be performed 2 ± 1 months after inclusion and will consist of a clinical evaluation, echocardiography, 24-hour Holter, or prolonged electrocardiographic monitoring (data collection form - Appendix B). A complete and integrated genotype-phenotype analysis of the cases included will be performed. Patients and their families will be followed for a minimum of 2 years and a maximum of 5 years and they will be evaluated annually with clinical consultations and with the same complementary methods described above.

PROCEDURES Collection and purification of DNA samples Genomic DNA will be purified from peripheral blood or mouth swabs. Whole blood will be collected by peripheral phlebotomy in tubes containing K2EDTA as an anticoagulant. Blood samples will be stored at 4-8 oC for up to a week before DNA purification. Mouth swabs will be collected using the ORAcollect • DNA kit (OCR-100) (DNA Genotek Inc., Canada). Genomic DNA from whole blood or mouth swab samples will be purified using DNeasy Blood & Tissue Kit (QIAGEN).

The analysis of germline genetic variants (inherited or de novo) through DNA sequencing, either by the Sanger method or by new generation sequencing, is not influenced by the tissue or body fluid from which the DNA is purified. Therefore, peripheral blood or oral smears/saliva can be used as a source of DNA without any technical compromise or introduction of bias. Thus, the choice of blood or oral swab will be determined essentially by the comfort and convenience for the research participant and aiming at the rational use of the available resources.

DNA quantification and quality control The purified genomic DNA will be quantified by ultraviolet spectrophotometry using the NanoDrop microvolume spectrophotometer (ThermoFisher Scientific). DNA integrity will be measured by agarose gel electrophoresis and using the Agilent 4200 TapeStation system.

Genetic analysis strategy In the initial discovery phase, 20 probands will be selected for analysis of sequence and copy number variants within a panel of selected candidate genes. The suspicious causal variables identified in this initial phase will later be analyzed in up to 4 family members or first-degree relatives for each proband.

Genetic panel and gene selection criteria Candidate genes included in the panel were selected from searches in the Online Mendelian Inheritance in Man (OMIM) database, by reviewing the literature and consensus, recommendations, and guidelines issued by panels and specialist societies. The final list of candidate genes was established to include clinically informative genes, i.e., which assist in diagnostic or therapeutic decisions, and experimental evidence indicative of genetic involvement in the pathophysiology of arrhythmias.

New generation sequencing Candidate genes will be analyzed for the detection of sequence and copy number variants using new generation sequencing. The entire coding region and intron-exon boundaries will be sequenced using Ampliseq ™ technology. The oligonucleotides for the amplification of the regions of interest will be designed using the online tool Ion AmpliSeq Designer. The sequencing libraries will be generated using the Ion AmpliSeq ™ Library Kit on the Ion OneTouch 2 System (ThermoFisher Scientific). The sequencing will be performed on an Ion Personal Genome Machine (PGM) sequencer using the Ion 318 ™ Chip v2 BC and the Ion PGM ™ Hi-Q ™ View Sequencing reagents (ThermoFisher Scientific). Sequencing analysis will be performed using the Ion Reporter ™ software (ThermoFisher Scientific).

Interpretation and reporting of sequence variants. The interpretation and registration of sequence variants will be performed according to the consensual recommendation of the American College of Medical Genetics and Genomics, the Association for Molecular Pathology, and the College of American Pathologists. Briefly, to describe variants identified in genes that cause Mendelian disorders, this consensus recommends the use of standard terms: pathogenic, probably pathogenic, uncertain meaning, likely benign and benign. According to this recommendation, the process of classifying variants in these five categories is based on a series of different types of evidence, such as population data, computer simulations, functional data, and genetic segregation data.

The evaluation of the pathogenicity of the genetic variants that are detected will be done independently, i.e., "blind", by the specialists. The clinical evaluation of the patients and determination of the phenotype will be carried out by the arrhythmia specialists in the group under the supervision of Dr. Nilson Araújo. The genetic evaluation will be done in a 'blind' way by Dr. Marcelo Reis. In case of divergence between the variant found and the phenotype, the findings will be reviewed by Dr. Luciana Sacilotto (specialist in arrhythmia with experience in clinical genetics) and by Dr. Carolina Bustamante (specialist in molecular genetics).

Computational prediction of the functional effect of genetic variants To estimate the functional effects of the sequence variants, a series of publicly available tools will be used. These algorithms consider the evolutionary conservation of amino acid residues and conserved protein domains, protein structure and function, Hiden Markov models, and position-dependent logic. Whenever available, functional experimental data in vitro on the effect of specific sequence variants will also be considered for interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Rede D'or São Luiz and their relatives
* Patients whit arrhythmia and their relatives
* Presence of inheritance pattern of causal genetic variants or those associated with phenotypes jointly defined as cardiac channelopathies and their relatives

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients and family members accompanied by the arrhythmia group of Rede D'Or, Rio de Janeiro, Brazil. The number of individuals we intend to include in the study refers to a convenience sample based on patients currently followed by the group of specialists from Rede D'Or who are part of the study and their families. The choice of up to 4 family members per proband is justified by the fact that this number of related individuals is, in most cases, sufficient to determine the pattern of occurrence and segregation of phenotypes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
phenotypic analysis | Patients and their families will be followed up to 5 years
  by genomic DNA purified from peripheral blood or mouth swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Nilson O Araujo, Dr, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abriel H, Zaklyazminskaya EV. Cardiac channelopathies: genetic and molecular mechanisms. Gene. 2013 Mar 15;517(1):1-11. doi: 10.1016/j.gene.2012.12.061. Epub 2012 Dec 22. PMID 23266818
- [Result] Ackerman MJ, Priori SG, Willems S, Berul C, Brugada R, Calkins H, Camm AJ, Ellinor PT, Gollob M, Hamilton R, Hershberger RE, Judge DP, Le Marec H, McKenna WJ, Schulze-Bahr E, Semsarian C, Towbin JA, Watkins H, Wilde A, Wolpert C, Zipes DP; Heart Rhythm Society (HRS); European Heart Rhythm Association (EHRA). HRS/EHRA expert consensus statement on the state of genetic testing for the channelopathies and cardiomyopathies: this document was developed as a partnership between the Heart Rhythm Society (HRS) and the European Heart Rhythm Association (EHRA). Europace. 2011 Aug;13(8):1077-109. doi: 10.1093/europace/eur245. No abstract available. Erratum In: Europace. 2012 Feb;14(2):277. Probst, Vincent [added]; Schwartz, Peter J [added]; Kaab, Stefan [added]; Kirchhof, Paulus [added]. PMID 21810866
- [Result] Antzelevitch C, Brugada P, Borggrefe M, Brugada J, Brugada R, Corrado D, Gussak I, LeMarec H, Nademanee K, Perez Riera AR, Shimizu W, Schulze-Bahr E, Tan H, Wilde A. Brugada syndrome: report of the second consensus conference. Heart Rhythm. 2005 Apr;2(4):429-40. doi: 10.1016/j.hrthm.2005.01.005. PMID 15898165
- [Result] Bezzerides VJ, Zhang D, Pu WT. Modeling Inherited Arrhythmia Disorders Using Induced Pluripotent Stem Cell-Derived Cardiomyocytes. Circ J. 2016 Dec 22;81(1):12-21. doi: 10.1253/circj.CJ-16-1113. Epub 2016 Dec 3. PMID 27916777
- [Result] Brugada P, Brugada R, Brugada J. Should patients with an asymptomatic Brugada electrocardiogram undergo pharmacological and electrophysiological testing? Circulation. 2005 Jul 12;112(2):279-92; discussion 279-92. doi: 10.1161/CIRCULATIONAHA.104.485326. No abstract available. PMID 16009809
- [Result] Chugh SS, Huertas-Vazquez A. Inherited arrhythmia syndromes: exome sequencing opens a new door to diagnosis. J Am Coll Cardiol. 2014 Jan 28;63(3):267-8. doi: 10.1016/j.jacc.2013.07.089. Epub 2013 Sep 25. No abstract available. PMID 24076289
- [Result] Coumel P, Fidelle J, Lucet V, et al. Catecholamine-induced severe ventricular arrhythmias with Adams-Stokes syndrome in children: report of four cases. Br Heart J 1978;40(Suppl):28-37
- [Result] Fernandez-Falgueras A, Sarquella-Brugada G, Brugada J, Brugada R, Campuzano O. Cardiac Channelopathies and Sudden Death: Recent Clinical and Genetic Advances. Biology (Basel). 2017 Jan 29;6(1):7. doi: 10.3390/biology6010007. PMID 28146053
- [Result] Giudicessi JR, Ackerman MJ. Determinants of incomplete penetrance and variable expressivity in heritable cardiac arrhythmia syndromes. Transl Res. 2013 Jan;161(1):1-14. doi: 10.1016/j.trsl.2012.08.005. Epub 2012 Sep 17. PMID 22995932
- [Result] Giudicessi JR, Ackerman MJ. Genetic testing in heritable cardiac arrhythmia syndromes: differentiating pathogenic mutations from background genetic noise. Curr Opin Cardiol. 2013 Jan;28(1):63-71. doi: 10.1097/HCO.0b013e32835b0a41. PMID 23128497
- [Result] Gollob MH, Blier L, Brugada R, Champagne J, Chauhan V, Connors S, Gardner M, Green MS, Gow R, Hamilton R, Harris L, Healey JS, Hodgkinson K, Honeywell C, Kantoch M, Kirsh J, Krahn A, Mullen M, Parkash R, Redfearn D, Rutberg J, Sanatani S, Woo A. Recommendations for the use of genetic testing in the clinical evaluation of inherited cardiac arrhythmias associated with sudden cardiac death: Canadian Cardiovascular Society/Canadian Heart Rhythm Society joint position paper. Can J Cardiol. 2011 Mar-Apr;27(2):232-45. doi: 10.1016/j.cjca.2010.12.078. PMID 21459272
- [Result] Hofman N, Tan HL, Alders M, van Langen IM, Wilde AA. Active cascade screening in primary inherited arrhythmia syndromes: does it lead to prophylactic treatment? J Am Coll Cardiol. 2010 Jun 8;55(23):2570-6. doi: 10.1016/j.jacc.2009.12.063. PMID 20513597
- [Result] Ingles J, Zodgekar PR, Yeates L, Macciocca I, Semsarian C, Fatkin D; CSANZ Cardiac Genetic Diseases Council Writing Group. Guidelines for genetic testing of inherited cardiac disorders. Heart Lung Circ. 2011 Nov;20(11):681-7. doi: 10.1016/j.hlc.2011.07.013. PMID 22000298
- [Result] Li MM, Datto M, Duncavage EJ, Kulkarni S, Lindeman NI, Roy S, Tsimberidou AM, Vnencak-Jones CL, Wolff DJ, Younes A, Nikiforova MN. Standards and Guidelines for the Interpretation and Reporting of Sequence Variants in Cancer: A Joint Consensus Recommendation of the Association for Molecular Pathology, American Society of Clinical Oncology, and College of American Pathologists. J Mol Diagn. 2017 Jan;19(1):4-23. doi: 10.1016/j.jmoldx.2016.10.002. PMID 27993330
- [Result] Medeiros-Domingo A, Bhuiyan ZA, Tester DJ, Hofman N, Bikker H, van Tintelen JP, Mannens MM, Wilde AA, Ackerman MJ. The RYR2-encoded ryanodine receptor/calcium release channel in patients diagnosed previously with either catecholaminergic polymorphic ventricular tachycardia or genotype negative, exercise-induced long QT syndrome: a comprehensive open reading frame mutational analysis. J Am Coll Cardiol. 2009 Nov 24;54(22):2065-74. doi: 10.1016/j.jacc.2009.08.022. PMID 19926015
- [Result] Mizusawa Y, Wilde AA. Brugada syndrome. Circ Arrhythm Electrophysiol. 2012 Jun 1;5(3):606-16. doi: 10.1161/CIRCEP.111.964577. No abstract available. PMID 22715240
- [Result] Nademanee K, Veerakul G, Chandanamattha P, Chaothawee L, Ariyachaipanich A, Jirasirirojanakorn K, Likittanasombat K, Bhuripanyo K, Ngarmukos T. Prevention of ventricular fibrillation episodes in Brugada syndrome by catheter ablation over the anterior right ventricular outflow tract epicardium. Circulation. 2011 Mar 29;123(12):1270-9. doi: 10.1161/CIRCULATIONAHA.110.972612. Epub 2011 Mar 14. PMID 21403098
- [Result] Priori SG, Wilde AA, Horie M, Cho Y, Behr ER, Berul C, Blom N, Brugada J, Chiang CE, Huikuri H, Kannankeril P, Krahn A, Leenhardt A, Moss A, Schwartz PJ, Shimizu W, Tomaselli G, Tracy C; Document Reviewers; Ackerman M, Belhassen B, Estes NA 3rd, Fatkin D, Kalman J, Kaufman E, Kirchhof P, Schulze-Bahr E, Wolpert C, Vohra J, Refaat M, Etheridge SP, Campbell RM, Martin ET, Quek SC; Heart Rhythm Society; European Heart Rhythm Association; Asia Pacific Heart Rhythm Society. Executive summary: HRS/EHRA/APHRS expert consensus statement on the diagnosis and management of patients with inherited primary arrhythmia syndromes. Europace. 2013 Oct;15(10):1389-406. doi: 10.1093/europace/eut272. Epub 2013 Aug 30. No abstract available. PMID 23994779
- [Result] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Result] Schwartz PJ, Priori SG, Spazzolini C, Moss AJ, Vincent GM, Napolitano C, Denjoy I, Guicheney P, Breithardt G, Keating MT, Towbin JA, Beggs AH, Brink P, Wilde AA, Toivonen L, Zareba W, Robinson JL, Timothy KW, Corfield V, Wattanasirichaigoon D, Corbett C, Haverkamp W, Schulze-Bahr E, Lehmann MH, Schwartz K, Coumel P, Bloise R. Genotype-phenotype correlation in the long-QT syndrome: gene-specific triggers for life-threatening arrhythmias. Circulation. 2001 Jan 2;103(1):89-95. doi: 10.1161/01.cir.103.1.89. PMID 11136691
- [Result] Splawski I, Timothy KW, Sharpe LM, Decher N, Kumar P, Bloise R, Napolitano C, Schwartz PJ, Joseph RM, Condouris K, Tager-Flusberg H, Priori SG, Sanguinetti MC, Keating MT. Ca(V)1.2 calcium channel dysfunction causes a multisystem disorder including arrhythmia and autism. Cell. 2004 Oct 1;119(1):19-31. doi: 10.1016/j.cell.2004.09.011. PMID 15454078
- [Result] Wang Q, Shen J, Splawski I, Atkinson D, Li Z, Robinson JL, Moss AJ, Towbin JA, Keating MT. SCN5A mutations associated with an inherited cardiac arrhythmia, long QT syndrome. Cell. 1995 Mar 10;80(5):805-11. doi: 10.1016/0092-8674(95)90359-3. PMID 7889574
- [Result] Zellerhoff S, Pistulli R, Monnig G, Hinterseer M, Beckmann BM, Kobe J, Steinbeck G, Kaab S, Haverkamp W, Fabritz L, Gradaus R, Breithardt G, Schulze-Bahr E, Bocker D, Kirchhof P. Atrial Arrhythmias in long-QT syndrome under daily life conditions: a nested case control study. J Cardiovasc Electrophysiol. 2009 Apr;20(4):401-7. doi: 10.1111/j.1540-8167.2008.01339.x. Epub 2008 Oct 27. PMID 19017345